CLINICAL TRIAL: NCT07170735
Title: Quantitative Measurement of Plasma and Urine MTB Cell-free DNA Level in Diagnosing TB and Treatment Monitoring
Brief Title: Quantitative Measurement of Plasma and Urine MTB Cell-free DNA Level
Acronym: LIQUID-TB
Status: Not yet recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Ka Pang Chan, Assistant Professor, Chinese University of Hong Kong
Other Study IDs: LIQUID-MTB
Record Dates: First submitted 2025-09-05; First posted 2025-09-12 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Tuberculosis
Keywords: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Blood and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- TB group: patients with active TB disease
  Interventions: Diagnostic Test: Plasma MTB cfDNA assay; Diagnostic Test: Urine MTB cfDNA assay
- LTBI group: patients with latent TB infection
  Interventions: Diagnostic Test: Plasma MTB cfDNA assay; Diagnostic Test: Urine MTB cfDNA assay
- control group: subjects without active TB disease or latent TB infection
  Interventions: Diagnostic Test: Plasma MTB cfDNA assay; Diagnostic Test: Urine MTB cfDNA assay

INTERVENTIONS:
Diagnostic Test: Plasma MTB cfDNA assay — Quantitative measurement of MTB cfDNA level in the plasma
Diagnostic Test: Urine MTB cfDNA assay — Quantitative measurement of MTB cfDNA level in the urine

SUMMARY:
Tuberculosis (TB) is one of the leading causes of infectious disease worldwide. The diagnosis of TB typically relies on microbiological evidence of the presence of Mycobacterium tuberculosis (MTB) or histological features of the host immune response to MTB in the infected organs. The diagnosis can be enhanced by performing molecular diagnostic tests (e.g. polymerase chain reaction, PCR) on the clinical specimens obtained. Expectorated sputum is usually the first sample sent for MTB culture for suspected pulmonary TB (PTB), which is the most common type of TB. However, this can be particularly challenging for paediatric patients and elderly patients with poor coughing techniques or effort. While for extrapulmonary TB (EPTB), which contributes to 10-20% of TB cases, with TB pleuritis and lymphadenitis as the most common types, invasive investigations are usually required for obtaining clinical specimens of good quality for MTB culture or histological examination. The invasiveness of procedures (e.g. pleural biopsy, lymph node biopsy) and inadequate sensitivity of diagnostic tests could hinder the diagnosis of EPTB. The long turnaround time of MTB culture also creates a challenge for timely diagnosis. Blood sampling for MTB culture or PCR, although non-invasive, has low diagnostic yields. All these urges for non-invasive, rapid and accurate diagnosis of TB.

The standard duration of TB treatment is 6 months, with a longer duration up to 12 months required for certain types of EPTB or in patients with underlying comorbidities (e.g. diabetes mellitus). Treatment monitoring and surveillance for relapses are typically based on a composite of clinical symptoms, sputum MTB culture status, and radiographical appearance. All these domains have their drawbacks, including subjective reporting (clinical symptoms), long turnaround times (sputum MTB culture status), and a lack of diagnostic sensitivity (changes in radiographical appearance in PTB). These clinical unmet needs may be overcome if a non-invasive molecular test could accurately quantify the burden of MTB in the body. Recently, it was reported that the level of MTB cfDNA in plasma can be measured by the CRISPR-TB assay. However, the data were derived mainly from the paediatric patient group and did not evaluate the possibility of latent TB infection (LTBI). This new technology remains explorative at the moment.

Our group has developed a metagenomic sequencing-based assay for measuring the level of MTB cell-free DNA (cfDNA) in plasma. We hypothesize that this new plasma MTB cfDNA assay has the potential to diagnose active TB disease, treatment monitoring and surveillance monitoring by serially measuring the MTB cfDNA level in the plasma. Similar technology may also be applicable to urine, which requires prospective validation.

ELIGIBILITY:
Inclusion Criteria:

* TB group: patients hospitalized for newly diagnosed TB disease.
* LTBI group: patients without TB disease, but with LTBI diagnosed by either tuberculin skin test (TST) or an interferon-gamma release assay (IGRA) blood test.
* Control group: patients or healthy volunteers without TB disease and LTBI

Exclusion Criteria:

* History of prior TB disease.
* Concomitant use of at least two first-line anti-TB drugs for at least 2 weeks in the past 3 months.
* Aged 17 years or younger
* Life expectancy of less than 12 months
* Failed to obtain informed consent due to the patient's refusal or cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with active TB disease will be recruited as positive control. Patients with latent TB infection, and subjects without active TB disease and latent TB infection will be recruited as negative control.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
diagnostic performance of the plasma MTB cfDNA assay | 1 month
  The diagnostic performance of the plasma MTB cfDNA assay in patients with newly diagnosed TB disease

SECONDARY OUTCOMES:
Level of plasma MTB cfDNA level during treatment | 6 months
  Quantitative measurement of MTB cfDNA level during the course of anti-tuberculous treatment
Level of plasma MTB cfDNA level after treatment | 3 months
  Quantitative measurement of MTB cfDNA level after completing the anti-tuberculous treatment
diagnostic performance of the urine MTB cfDNA assay | 1 month
  The diagnostic performance of the urine MTB cfDNA assay in patients with newly diagnosed TB disease
Level of urine MTB cfDNA level during treatment | 6 months
  Quantitative measurement of MTB cfDNA level during the course of anti-tuberculous treatment
Level of urine MTB cfDNA level after treatment | 3 months
  Quantitative measurement of MTB cfDNA level after completing the anti-tuberculous treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No